CLINICAL TRIAL: NCT06268158
Title: The Effect of Eye Mask and Music on Sleep Quality and Delirium in Patients Monitored in Intensive Care Unit Following Abdominal Surgery
Brief Title: The Effect of Eye Mask and Music on Sleep Quality and Delirium in Patients Monitored in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yeliz Sürme, Assoc.Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/45
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Surgery
Keywords: abdominal surgery; delirium; sleep quality; eye patch; music
MeSH Terms: conditions — Delirium; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the experimental group will wear an eye patch after 22:00, when clinical interventions are less frequent, and will be listened to calming music once a day for 1 hour for 3 days.
  Interventions: Behavioral: Eye patch
- Control group (No Intervention): No treatment will be performed on patients in the control group outside of their clinical routine.

INTERVENTIONS:
Behavioral: Eye patch — The experimental group will fill out the patient introduction form, Richmond Agitation-Sedation Scale, Nursing Delirium Screening Scale and Richard-Campbell Sleep Scale on the first day. On the 4th day of the study, the Nursing Delirium Screening Scale and the Richard-Campbell Sleep Scale will be completed.
  Other Names: Music
  Arms: Intervention group

SUMMARY:
After abdominal surgery, most patients experience problems such as respiratory complications, surgical wound infection, cardiac problems, renal failure, delirium, and insomnia, along with surgical trauma and underlying comorbidities. Postoperative delirium (POD) is an adverse postoperative complication that can occur in patients of all ages, from children to the elderly. Effective non-pharmacological treatment approaches for delirium include using an orientation board, calendar, clock, ensuring hydration, improving sleep quality, therapeutic activities, providing companionship of family members, and building private rooms. This study conducted as a randomized controlled and experimental study to determine the effect of eye patch and music on sleep quality and delirium in patients followed after abdominal surgery in the surgical intensive care unit.

It was planned to include a total of 34 patients who underwent abdominal surgery, 17 in the experimental group and 17 in the control group.Considering possible sample loss, the study was completed with 45 patients, 21 in the experimental group and 24 in the control group.

During the data collection phase, the Patient Information Form, Richard-Campbell Sleep Scale, Nursing Delirium Screening Scale and Richmond Agitation-Sedation Scale, were used.

ELIGIBILITY:
Inclusion Criteria:

* Those who have had abdominal surgery
* Those who volunteer to participate in the research
* Those who are over 18 years old
* Richmond Agitation-Sedation Scale -1, 0, +1
* Those who have been in intensive care for at least 3 days
* No communication problems (language, hearing impairment, etc.)
* No mental problems
* Patients who do not use sleeping pills or sedating drugs and who do not have alcohol or substance addiction will be included in the study.

Exclusion Criteria:

* Those who experience blood loss and fluid electrolyte imbalance after surgery
* There are contraindications to the use of eye masks (for example, head trauma),
* Patients with delirium before or after surgery will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Richard-Campbell Sleep Scale | day 1 and 4 of the study
  It is a scale consisting of 6 items that evaluate the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake when waking up, the quality of sleep and the noise level in the environment. The 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation.
  Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep.
Nursing Delirium Screening Scale | day 1 and 4 of the study
  The scale consists of 5 items, including disorientation, inappropriate behavior, inappropriate communication, illusion-hallucination and slowing down of psychomotor behaviors. Each item in the scale receives a value between 0 and 2 points, and the total score varies between 0 and 10. A score of two and above indicates delirium.

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale | day 1
  It is a 10-point scale with four levels indicating anxiety and agitation (1-4), one level indicating calm and alertness (0), and five levels indicating sedation stages (-1;-5). Richmond agitation sedation scale scores range from +4 to -5. Positive RASS scores indicate agitated patients, negative scores indicate sedated or comatose patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Sürme, PhD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puppo Moreno AM, Abella Alvarez A, Morales Conde S, Perez Flecha M, Garcia Urena MA. The intensive care unit in the postoperative period of major abdominal surgery. Med Intensiva (Engl Ed). 2019 Dec;43(9):569-577. doi: 10.1016/j.medin.2019.05.007. Epub 2019 Aug 1. English, Spanish. PMID 31377023
- [Background] Linke GR, Mieth M, Hofer S, Trierweiler-Hauke B, Weitz J, Martin E, Buchler MW. Surgical intensive care unit - essential for good outcome in major abdominal surgery? Langenbecks Arch Surg. 2011 Apr;396(4):417-28. doi: 10.1007/s00423-011-0758-y. Epub 2011 Mar 3. PMID 21369847
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743